CLINICAL TRIAL: NCT05431374
Title: A Randomized Controlled Trial of Measurement-Based Care Vs. Standard Care for Major Depressive Disorder in Pakistan
Brief Title: Measurement-Based Care Vs. Standard Care for Major Depressive Disorder
Acronym: MBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBC-Depression; Depression (Other: PILL)
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Measurement Based Care MBC; Pakistan
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 allocation to measurement-based vs. standard-care.
Who Masked: Outcomes Assessor
Masking Description: This will be an assessor blind, randomized controlled trial. Due to the nature of the interventions, it will be impossible to blind clinicians in participating centres or the participants themselves. Before assessments, participants will be asked not to reveal any information about treatment to assessors. To avoid unblinding, outcome assessors will be located separately from treatment providers, and we will assign new outcome assessors in cases of unintentional unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Measurement Based Care MBC (Experimental): patients in the MBC group will receive treatment according to a schedule that includes individualized starting dosages, dosage adjustment, and medication changes to minimize side effects, maximize safety, and optimize the therapeutic benefit for each patient.
  Interventions: Other: Measurement Based Care (MBC)
- Control/Standard-care (Active Comparator): Local medical, psychiatric and family medicine services provide routine care according to their clinical judgment and available resources. Standard-care will be ascertained by the participant's treating physician. Research staff will record the nature and intensity of standard-care delivered to each participant. In current practice, MDD patients are not routinely referred for any psychological therapies in Pakistan. Standard-care in Pakistan largely comprises of pharmacotherapy.
  Interventions: Other: Control/Standard-care

INTERVENTIONS:
Other: Measurement Based Care (MBC) — Patients in both groups will receive either open-label paroxetine (10-40mg/day) or open-label mirtazapine (7.5-45mg/day), within the therapeutic dosage range recommended by the US Food and Drug Authority (Paxil -Highlights of Prescribing Medication, 2022; Remeron -Highlights of Prescribing Medication, 2022). Paroxetine, a selective serotonin reuptake inhibitor, is chosen because it has been one of the most commonly prescribed antidepressants, and mirtazapine, an alpha-2 antagonist, is chosen because it has a different mechanism of action. The treating psychiatrists will decide which of the antidepressants and dosages to prescribe, as long as they were within the study's recommended dosage ranges.
  patients in the MBC group will receive treatment according to a schedule that includes individualized starting dosages, dosage adjustment, and medication changes to minimize side effects, maximize safety, and optimize the therapeutic benefit for each patient.
  Arms: Measurement Based Care MBC
Other: Control/Standard-care — Local medical, psychiatric and family medicine services provide routine care according to their clinical judgment and available resources. Standard-care will be ascertained by the participant's treating physician. Research staff will record the nature and intensity of standard-care delivered to each participant. In current practice, MDD patients are not routinely referred for any psychological therapies in Pakistan. Standard-care in Pakistan largely comprises of pharmacotherapy.
  Arms: Control/Standard-care

SUMMARY:
Major depressive disorder (MDD) is one of the leading causes of disability worldwide, indicated as one of the two most disabling mental disorders by the Global Burden of Diseases, Injuries, and Risk Factors Study (GBD) 2019 (Vos et al., 2020). Despite several effective pharmacological and psychosocial interventions available globally, only about one-third of depressed patients achieve remission (Xiao et al., 2021). There is a need to establish scalable clinical management practices which utilize biopsychosocial assessments, formulate a differential diagnosis, and provide evidence-based treatments for patients with MDD (Hong et al., 2021). While significant evidence for effectiveness of Measurement Based Care (MBC) is found in clinical settings from high and middle-income countries, assessments of MBC compared with usual care for the treatment of MDD are yet to be completed in low-resource settings like LMICs. The aim of this trial is to determine the efficacy and safety of MBC in patients with MDD in comparison with standard care in Pakistan. In order to reduce the variance found in treatment-as-usual and isolate the impact of MBC, standard care for this trial will limit medication choices to either paroxetine or mirtazapine.

DETAILED DESCRIPTION:
Hypothesis: The rates of response and remission, and time to response and remission would be significantly shorter in the MBC group, without greater dropout rates and side effect burden, compared with the standard treatment group.

Study design and setting This will be a multi-centre, with assessors blind to protocol and treatment group, parallel arm, randomized controlled trial (RCT). The study is a direct replication of a study conducted by Gou et al. (2015) in China.

Participants Participants will be recruited from psychiatric units of teaching and non-teaching hospitals in 6 centres: Karachi (population 23 million), Lahore (population 10 million), Rawalpindi (population 3 million), Hyderabad (population 2 million) and Quetta (population 1 million) and Multan (1.8 million).

Sample size The sample size of 120 participants for this exploratory trial is based on the study conducted by Guo et al.

ELIGIBILITY:
Inclusion Criteria:

1. Adult outpatients age 18-65 of age
2. Diagnosis of nonpsychotic MDD established by treating psychiatrists and confirmed by a checklist based on DSM-5 criteria at study entry
3. Currently depressed with a score >17 on the 17-item Hamilton Depression Rating (HDRS-17)
4. Able to communicate effectively and give written informed consent
5. Resident of the trial catchment area.

Exclusion Criteria:

1. Lifetime history of drug or alcohol dependence; 2. Diagnosis of bipolar, psychotic, obsessive-compulsive, or eating disorders confirmed with DSM-5 criteria 3. History of a lack of response or intolerance to either of the two protocol antidepressants (paroxetine and mirtazapine) 4. Currently pregnancy or breastfeeding; 5. Suicide attempts in the current depressive episode; 6. Any major medical condition contraindicating the use of the protocol antidepressants.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating (HDRS-17) - Time to Response | Time from baseline to response (in weeks) (assessed upto 24 weeks).
  is a 17-item instrument that was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Ratings are made using either a five- or a three-point scale, yielding total scores from zero to 61. Response will be defined as a decrease of 50% from the baseline HDRS-17 score.
Hamilton Depression Rating (HDRS-17) - Time to Remission | Time from baseline to remission (in weeks) (assessed upto 24 weeks)
  is a 17-item instrument that was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Ratings are made using either a five- or a three-point scale, yielding total scores from zero to 61. Remission as a HDRS-17 score<7

SECONDARY OUTCOMES:
Hamilton Depression Rating (HDRS-17) - Severity | Change in scores from baseline to 3-month and 6-month follow up
  is a 17-item instrument that was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Ratings are made using either a five- or a three-point scale, yielding total scores from zero to 61. Higher scores indicate higher severity.
Adverse Effect Checklist | Rates of adverse effects from baseline to 6-month follow up
  This checklist includes some common adverse effects of antidepressant medications.
All-cause discontinuation | Time from baseline to all-cause discontinuation of antidepressant medication (assessed upto 24 weeks)
  Discontinuation from participation in the study.

CONTACTS AND LOCATIONS:
Locations (6):
- Pakistan (6):
  - Bolan Medical Complex, Quetta, Balochistan
  - Services Hospital, Lahore, Punjab Province
  - Nishtar Hospital, Multan Khurd, Punjab Province
  - Benazir Bhutto Hospital, Rawalpindi, Punjab Province
  - Civil Hospital, Karachi, Sindh
  - Civil Hospital, Hyderābād

IPD SHARING:
Plan to Share IPD: No
Only anonymized data will be shared with researchers

REFERENCES:
- [Derived] Husain MI, Nigah Z, Ansari SUH, Khoso AB, Kiran T, Umer M, Ansari MA, Bhatia MR, Khan SA, Husain MO, Malik AG, Naqvi HA, Qadir A, Rajput AH, Saqib M, Ilyas M, Doutani MUK, Sherzad S, Siddiqui KMS, Tahir Z, Wang W, Husain N, Chaudhry N, Chaudhry IB, Mulsant BH. Measurement-Based Care to Enhance Antidepressant Treatment Outcomes in Major Depressive Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2529427. doi: 10.1001/jamanetworkopen.2025.29427. PMID 40892412